CLINICAL TRIAL: NCT02759796
Title: Indocyanine Green Fluorescence Angiography in the Assessment of Deep Inferior Epigastric Perforator (DIEP) Flap Perfusion
Brief Title: Fluorescence Angiography in the Assessment of DIEP Flap Perfusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: idipaz
Record Dates: First submitted 2016-04-05; First posted 2016-05-03 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Breast Cancer; Vascularization; Fat Necrosis
MeSH Terms: conditions — Breast Neoplasms; Neovascularization, Pathologic; Fat Necrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clinical assessment of flap perfusion (Placebo Comparator): Tailoring the flap according to clinical assessment of flap perfusion
  Interventions: Procedure: Tailoring the flap according to clinical assessment
- Angiography assessment of flap perfusion (Experimental): Tailoring the flap according to ICG Angiography assessment of flap perfusion
  Interventions: Procedure: Tailoring the flap according to ICG Angiography assessment

INTERVENTIONS:
Procedure: Tailoring the flap according to clinical assessment — After microvascular anastomosis is performed, the investigators clinically assess flap vascularization and the well vascularized tissue is marked by means of a dermographic pencil. Then the investigators administer 0,2mg/kg of ICG intravenously. The vascularization of the flap is also checked by means of the Photo Dynamic Eye (Pulsion Medical System) but finally the decision of discarding the poorly vascularized areas of the flap is made by clinical assessment.
  Arms: Clinical assessment of flap perfusion
Procedure: Tailoring the flap according to ICG Angiography assessment — After microvascular anastomosis is performed, the investigators administer 0,2mg/kg of ICG intravenously. Then the investigators check the vascularization of the flap by means of the Photo Dynamic Eye (Pulsion Medical System) and the poorly vascularized areas of the flap are discarded guided by ICG perfusion test.
  Arms: Angiography assessment of flap perfusion

SUMMARY:
It is a single-center, prospective, randomized and controlled study focused in microsurgical autologous breast reconstruction. It involves applying indocyanine green (ICG) angiography for the study of the vascularization of DIEP flaps. The aim of the study is to determine whether there are differences in complications and aesthetic results when ICG is used to discard the poorly vascularized areas of the flap. The study includes adult women undergoing unilateral DIEP flap breast reconstruction. The calculated sample size is 60 patients. There are two groups. In group 1, the investigators use the usual clinical criteria to discard the poorly vascularized areas of the flap. In group 2, the investigators use the ICG to shape the flap.

ELIGIBILITY:
Inclusion Criteria:

* Mastectomized adult female patient
* Abdominal flap unilateral breast reconstruction indication
* Alloplastic breast reconstruction sequelae
* Enough amount of abdominal dermofat tissue to shape a breast with a primary closure of the donor site

Exclusion Criteria:

* DIEP flap bilateral breast reconstruction indication
* Previous abdominoplasty surgery
* Untreated psychiatric disease
* Untreated infection
* Indocyanine green or iodine hypersensitivity
* Hyperthyroidism, thyroid adenoma or thyroid autonomy
* Any concomitant disease or condition that, in the opinion of the investigator, can make the patient unsuitable to receive a microsurgical technique or to join the research.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-11; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with fat necrosis as assessed by physical examination | Six months postoperatively
Number of participants with fat necrosis as assessed by ultrasonography | Six months postoperatively

SECONDARY OUTCOMES:
Number of participants with flap failure as assessed by physical examination | From intraoperative moment to one week postoperatively
Number of participants with wound infection as assessed by physical examination | From one day postoperatively to two weeks postoperatively
Number of participants with wound healing delay as assessed by physical examination | From two weeks postoperatively to two months postoperatively
Number of participants with reoperation | From immediate postoperative moment to one year postoperatively
Flap perfusion index as assessed by IC-CALC software (Pulsion Medical System) | Intraoperatively
Flap weight (grams) | Intraoperatively
Flap length (centimeters) | Intraoperatively
Breast-Q questionnaire (preoperative reconstruction module) to measure patient preoperative status | A preoperative test in the last week before surgery
Breast-Q questionnaire (postoperative reconstruction module) to measure patient postoperative status | A postoperative test one year after surgery
ICG security (Number of participants with tachycardia, exanthema and anaphylactic shock as assessed by physical examination and intraoperative monitoring) | Intraoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Luis Landín Jarillo, MD, PhD, Principal Investigator — La Paz University Hospital
Locations (1):
- La Paz University Hospital, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Varela R, Casado-Sanchez C, Zarbakhsh S, Diez J, Hernandez-Godoy J, Landin L. Outcomes of DIEP Flap and Fluorescent Angiography: A Randomized Controlled Clinical Trial. Plast Reconstr Surg. 2020 Jan;145(1):1-10. doi: 10.1097/PRS.0000000000006393. PMID 31577664